CLINICAL TRIAL: NCT03191344
Title: Extended Application of Intraoperative Parathyroid Scores System(IPSS) in Thyroidectomy
Acronym: IPSS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fujian Medical University (Other)
Responsible Party: Principal Investigator, Bo Wang,MD, MS, Fujian Medical University
Other Study IDs: IPSS
Record Dates: First submitted 2017-06-15; First posted 2017-06-19 (Actual); Last update posted 2018-09-18 (Actual); Status verified 2018-09

CONDITIONS: Intraoperative Parathyroid Scores System
Keywords: Intraoperative Parathyroid Scores System; total thyroidectomy; thyroid cancer; hypoparathyroidism; prediction
MeSH Terms: conditions — Thyroid Neoplasms; Hypoparathyroidism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- with IPSS record/IPSS: the surgoen use the IPSS in all thyroidectomy
  Interventions: Behavioral: with IPSS
- Traditionaldescription Group/TD: the surgoen without the IPSS，use Traditional description

INTERVENTIONS:
Behavioral: with IPSS — all patient in one group use IPSS to record the parathyroid status. the other group operation as ordinary. record the parathyroid status in verbal description
  Groups: with IPSS record/IPSS

SUMMARY:
after established the Intraoperative Parathyroid Scores System (IPSS) for thyroidectomy we further extented the clinical value of Intraoperative Parathyroid Scores System in Treatment decisions of calcium treatment time and improve recognition skills of parathyroid in Clinicians

DETAILED DESCRIPTION:
IPSS includes transplantation Parathyroid Scores and in situ Parathyroid Scores, the investigators will establish the Intraoperative Parathyroid Scores System by parathyroid size and Blood supply, and recording IPSS, according to certain rules. We expand IPSS, including the description of the location of parathyroid after postoperative.Parathyroid hormone and calcium were test in d0, d1, d14, d60 post operation. The correlation between Intraoperative Parathyroid Scores and PTH calcium were calculated, and ROC curve and logistic regression were tested for the prediction value.and after that we further evaluate the relationship Between IPSS and calcium supplement time.and Whether IPSS enhance ability of parathyroid recognition for clinical doctors.

ELIGIBILITY:
Inclusion Criteria:

1. postoperative pathology confirmed as thyroid papillary carcinoma;
2. for the first time to undergo thyroid surgery, no history of neck surgery and external radiotherapy;
3. preoperative serum calcium, parathyroid hormone levels were normal;
4. intraoperative and postoperative clinical data integrity, standardized follow-up patients;
5. parathyroid is a tumor violation.

Exclusion Criteria:

1. serious underlying disease;
2. age greater than 60 years of age or combined with arteriosclerotic disease;
3. patients with postoperative loss;
4. patients with parathyroid disease.

Max Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: the patients with thyroid tumors and require surgery In accordance with the guidelines.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2017-07-01 (Actual); Primary Completion 2019-07-01 (Estimated); Study Completion 2019-07-01 (Estimated)

PRIMARY OUTCOMES:
Differences of parathyroid records between IPSS and TD | 1 year
  The percentage of recorded integrity of the parathyroid gland and the number of recognizable parathyroids were compared between the two groups.

SECONDARY OUTCOMES:
The effect of IPSS on the level of parathyroid recognition of surgeons | 1 year
  Comparison of the number of parathyroid gland found in the pathology and the number of postoperative hypoparathyroidism between the two groups
differences of the number of parathyroid glands found in the pathology betwen IPSS and TD | 1 year
  differences of the number of parathyroid glands found in the pathology betwen IPSS and TD

OTHER OUTCOMES:
The Predictive Value of IPSS for Intravenous and Oral Calcium duration | 1 year
  Comparison of the correlation between IPSS values and intravenous calcium supplementation and oral calcium supplementation time.

CONTACTS AND LOCATIONS:
Locations (1):
- Wen-xin ZHAO, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No